CLINICAL TRIAL: NCT02265549
Title: Value of Radiomics for the Prediction of Long Term Survival and Local Failure After Stereotactic Radiotherapy (SRT) for Brain Metastases
Brief Title: Radiomics for Prediction of Long Term Survival and Local Failure After Stereotactic Radiotherapy for Brain Metastases
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: Radiomics SRT 09-2014
Record Dates: First submitted 2014-10-01; First posted 2014-10-16 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Metastases, Neoplasm
Keywords: Metastases,; Neoplasm; Cerebral
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Published prognostic scores have limitations in prediction of long term survival after stereotactic radiotherapy for brain metastases. Moreover, no validated tools are available for prediction of local failure. The value of radiomics is evaluated in this perspective.

DETAILED DESCRIPTION:
Sensitivity is low for prediction of long term survival of currently available prognostic scores for brain metastases. First the current clinical models will be optimized with a new prognostic model and nomogram. Radiomics is a tool to analyze tumor characteristics based on CT and MR images. These tumor characteristics may reflect tumor biology and outcome. Therefore it is investigated if radiomics improves prediction of long term survival after stereotactic radiotherapy for brain metastases. Moreover, the predictive value of radiomics for local failure is investigated.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral metastasized patients

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with 1 upto 4 brain metastases treated with SRT
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2014-09-04 (Actual); Study Completion 2014-09-04 (Actual)

PRIMARY OUTCOMES:
Sensitive value of 12 months survival after stereotactic radiotherapy for brain metastases with radiomics | 1 year
  Sensitivity of 12 months survival after stereotactic radiotherapy for brain metastases with radiomics. Radiomics is a tool to analyze tumor characteristics based on CT and MR images.
Sensitive value of 12 months local failure after stereotactic radiotherapy for brain metastases with radiomics | 1 year
  Sensitivity of 12 months local failure after stereotactic radiotherapy for brain metastases with radiomics. Radiomics is a tool to analyze tumor characteristics based on CT and MR images.

SECONDARY OUTCOMES:
Specificity of 12 months survival and local failure after stereotactic radiotherapy for brain metastases with radiomics. | 1 year
  Specificity of 12 months survival and local failure after stereotactic radiotherapy for brain metastases with radiomics.
Positive predictive value of 12 months survival and local failure after stereotactic radiotherapy for brain metastases with radiomics. | 1 year
  Positive predictive value of 12 months survival and local failure after stereotactic radiotherapy for brain metastases with radiomics.
Negative predictive value of 12 months survival and local failure after stereotactic radiotherapy for brain metastases with radiomics. | 1 year
  Negative predictive value of 12 months survival and local failure after stereotactic radiotherapy for brain metastases with radiomics.

OTHER OUTCOMES:
Area under the curve of published prognostic scores | 1 year
  Area under the curve published prognostic scores
Mismatch rate of published prognostic scores | 1 year
  Mismatch rate of published prognostic scores

CONTACTS AND LOCATIONS:
Locations (1):
- Maastro Clinic, Maastricht, Netherlands

REFERENCES:
- [Result] Zindler JD, Rodrigues G, Haasbeek CJ, De Haan PF, Meijer OW, Slotman BJ, Lagerwaard FJ. The clinical utility of prognostic scoring systems in patients with brain metastases treated with radiosurgery. Radiother Oncol. 2013 Mar;106(3):370-4. doi: 10.1016/j.radonc.2013.01.015. Epub 2013 Mar 20. PMID 23522151
- [Result] Rodrigues G, Zindler J, Warner A, Lagerwaard F. Recursive partitioning analysis for the prediction of stereotactic radiosurgery brain metastases lesion control. Oncologist. 2013;18(3):330-5. doi: 10.1634/theoncologist.2012-0316. Epub 2013 Feb 19. PMID 23429647
- [Result] Aerts HJ, Velazquez ER, Leijenaar RT, Parmar C, Grossmann P, Carvalho S, Bussink J, Monshouwer R, Haibe-Kains B, Rietveld D, Hoebers F, Rietbergen MM, Leemans CR, Dekker A, Quackenbush J, Gillies RJ, Lambin P. Decoding tumour phenotype by noninvasive imaging using a quantitative radiomics approach. Nat Commun. 2014 Jun 3;5:4006. doi: 10.1038/ncomms5006. PMID 24892406